CLINICAL TRIAL: NCT00031408
Title: Plan for Obtaining Informed Consent to Use Stored Human Biological Materials (HBM) for Currently Unspecified Analyses
Brief Title: Consent for Use of Stored Patient Specimens for Future Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5128; 1U01AI068636 (NIH)
Record Dates: First submitted 2002-03-05; First posted 2002-03-06 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: Specimen Handling; Blood; Informed Consent; Genetic Screening
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to obtain informed consent to use stored human biological materials (HBM) (e.g., blood and other tissues) for future studies that may include genetic testing.

DETAILED DESCRIPTION:
During past, present, and future Adult AIDS Clinical Trials Group (AACTG) clinical trials, samples of HBM (e.g., blood, other body fluids and tissues) have been or will be obtained and stored until analyzed, as defined by the particular trial for which the patient provided consent. Some HBM may be left over after a trial is completed. Important questions may arise during the design of a study; some of these questions may be addressed only with archived (rather than prospectively collected) HBMs. To improve understanding of HIV disease and its optimal management, it is critical that HBMs be available to investigators for subsequent unspecified analyses.

All patients are asked to sign the informed consent form and specify whether or not they agree to allow their leftover samples to be used for secondary analyses and whether or not they agree to have one 14 ml blood sample drawn in this study for DNA archiving for use in currently unspecified genetic analyses. Only under extraordinary circumstances will any individual patient from whom HBM was obtained be notified of any test result from secondary testing. Patients who do not agree to either option will indicate this on the informed consent and will have no further involvement in this study. Declining consent does not in any way jeopardize participation in any other current or future ACTG clinical trial. Consent may be obtained at the same time the patient is being enrolled into any ACTG clinical trial, at some interval after the patient has entered but is still participating in a trial, or at any time after the patient has completed participation in a trial. The goal of this study is to allow archived HBM to be used for research purposes while protecting the identity of patients from whom such samples were obtained. The focus is on obtaining permission to analyze archived HBM in ways not planned at the time the initial informed consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian willing to give informed consent, if applicable
* Either currently participating in or have ever participated in an AACTG clinical trial

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected individuals
Sampling Method: Non-Probability Sample
Enrollment: 17444 (Actual)
Dates: Start 2002-02-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Haas, MD, Study Chair — Vanderbilt University Medical Center
Locations (63):
- United States (62):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Charles Drew Medical Center, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Willow Clinic / Stanford Univ, Stanford, California
  - Harbor General/UCLA, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Department of Internal Medicine, University of Iowa Hospitals & Clinics CRS (1504), Iowa City, Iowa
  - Univ of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - Specialty Care Center CRS 1505, Omaha, Nebraska
  - New Jersey Medical School- Adult CRS (31477), Newark, New Jersey
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - The Cornell Clinical Trials Unit, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Community Health Network Inc, Rochester, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Wake County Health and Human Services CRS (30076), Chapel Hill, North Carolina
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic (A2508), Cleveland, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - The Research & Education Group-Portland CRS (31474), Portland, Oregon
  - Penn Therapeutics CRS (6201), Philadelphia, Pennsylvania
  - Presbyterian Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania, ACTU, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Dallas VA Medical Center (3752), Dallas, Texas
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS (31475), Richmond, Virginia
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Bronke C, Almeida CM, McKinnon E, Roberts SG, Keane NM, Chopra A, Carlson JM, Heckerman D, Mallal S, John M. HIV escape mutations occur preferentially at HLA-binding sites of CD8 T-cell epitopes. AIDS. 2013 Mar 27;27(6):899-905. doi: 10.1097/QAD.0b013e32835e1616. PMID 23276808